CLINICAL TRIAL: NCT06664723
Title: Effect of High Tone External Muscle Stimulation on Diabetic Foot Ulcer
Brief Title: High Tone External Muscle Stimulation on Diabetic Foot Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, PHD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005336
Record Dates: First submitted 2024-10-17; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: High tone; Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: high tone external muscle stimulation (Experimental): The study group will include 40 patients with diabetic foot ulcer receiving high tone external muscle stimulation three times a week for 8 weeks; in addition to Standard Medical Treatment: The Standard care of diabetic foot ulcers includes good glycemic control, adequate nutrition, off-loading (via bed rest or casts), local care (moist dressings and topical management), lessening of edema, surgical debridement of devitalized wound tissue and antibiotic therapy.
  Interventions: Device: high tone external muscle stimulation; Other: Standard medical treatment (SMT)
- Group B: Control (Sham Comparator): The control group will include 40 patients with diabetic foot ulcer receiving Standard Medical Treatment only. The Standard care of diabetic foot ulcers includes good glycemic control, adequate nutrition, off-loading (via bed rest or casts), local care (moist dressings and topical management), lessening of edema, surgical debridement of devitalized wound tissue and antibiotic therapy.
  Interventions: Other: Standard medical treatment (SMT)

INTERVENTIONS:
Device: high tone external muscle stimulation — Device HiToP®: Parameters of (HTEMS), Voltage: 230-V Pulse widths: ≤350 mA. Electrical Frequency: Frequencies continuously scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 m W. Intensity: the electrical stimulation will be adjusted to a pleasant level that will not produce any pain or discomfortable paraesthesia, Duration 30 minutes per session. Electrodes will be placed around ulcer. It will be introduced 3 times per week, for 8 weeks Prior to intervention, skin sensation will be assessed using warm water in a test-tube (temperature), pin prick (pain) and cotton wool (light touch) to ascertain the skin sensitivity
  Arms: Group A: high tone external muscle stimulation
Other: Standard medical treatment (SMT) — The Standard care of diabetic foot ulcers includes good glycemic control, adequate nutrition, off-loading (via bed rest or casts), local care (moist dressings and topical management), lessening of edema, surgical debridement of devitalized wound tissue and antibiotic therapy.

SUMMARY:
In this study 80 patients will be randomly assigned into two equal groups (40 patients for each group):

1. Group A: Experimental: (high tone external muscle stimulation for diabetic foot ulcer).

   The study group will include 40 patients with diabetic foot ulcer receiving high tone external muscle stimulation three times a week for 8 weeks; in addition to Standard Medical Treatment: The Standard care of diabetic foot ulcers includes good glycemic control, adequate nutrition, off-loading (via bed rest or casts), local care (moist dressings and topical management), lessening of edema, surgical debridement of devitalized wound tissue and antibiotic therapy.
2. Group B: Control: The control group will include 40 patients with diabetic foot ulcer receiving Standard Medical Treatment only. The Standard care of diabetic foot ulcers includes good glycemic control, adequate nutrition, off-loading (via bed rest or casts), local care (moist dressings and topical management), lessening of edema, surgical debridement of devitalized wound tissue and antibiotic therapy.

DETAILED DESCRIPTION:
1. Assessment measures and procedures:

   1- Wound Healing:

   1.a- Extent of wound: The wound will be measured using Image J, open source digital imaging software developed at the National Institutes of Health (NIH) to measure wound area of the target wound, in mm2 (the largest foot wound if multiple wounds are present). Image J software has been used specifically for the measurement of diabetic foot ulcers with very high inter- and intra-rater reliability (p=0.997 and 0.999 respectively). The wound will be traced on acetate paper using a fine permanent marker for use in Image J and a standard distance photograph of the wound will be taken to document wound bed characteristics after physician debridement to healthy granulating tissue or healthy bleeding tissue is reached. A completely healed wound has complete epithelialization (William et al., 2017).

   1.b-Direct measurement of volume using physiological saline: The wound will be covered with a sterile polyurethane film and then filled up with physiological saline injected using a needle that pierces the film. The quantity of saline corresponds to the wound volume. Wound volume measurements will be taken at baseline, after 4 weeks (midpoint) and after 8 weeks (HUMBERT et al., 2004).
2. Treatment procedures:

Device HiToP®: Parameters of (HTEMS), Voltage: 230-V Pulse widths: ≤350 mA. Electrical Frequency: Frequencies continuously scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 m W. Intensity: the electrical stimulation will be adjusted to a pleasant level that will not produce any pain or discomfortable paraesthesia, Duration 30 minutes per session. Electrodes will be placed around ulcer. It will be introduced 3 times per week, for 8 weeks Prior to intervention, skin sensation will be assessed using warm water in a test-tube (temperature), pin prick (pain) and cotton wool (light touch) to ascertain the skin sensitivity (Abdel Moez et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* - Male and female diabetic patients (controlled type II diabetes mellitus) categorized as having a chronic diabetic foot ulcer.
* Patients with unilateral or bilateral grade II (full thickness) diabetic foot ulcers according to Wagner's classification for diabetic foot disease and lasting longer than four months.
* Their ages will range from 45 to 65 years
* All participants will provide informed consent form giving agreement to participation and publication of the results of the study.
* All patients will receive the same medical care for treatment of diabetic foot ulcer and not receiving any physical therapy modalities before the study.

Exclusion Criteria:

* - Any pathological conditions or associated injuries affect the result of the study.
* Skin disease or any disease lead to ulcer other than diabetes as venous or arterial disease.
* Active malignancy and osteomyelitis associated with a diabetic foot ulcer.
* Any mental, cognitive and psychological impairment.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Extent of wound (wound surface area) | 8 weeks
  The wound will be measured using Image J, open source digital imaging software developed at the National Institutes of Health (NIH) to measure wound area of the target wound, in mm2 (the largest foot wound if multiple wounds are present). Image J software has been used specifically for the measurement of diabetic foot ulcers with very high inter- and intra-rater reliability (p=0.997 and 0.999 respectively). The wound will be traced on acetate paper using a fine permanent marker for use in Image J and a standard distance photograph of the wound will be taken to document wound bed characteristics after physician debridement to healthy granulating tissue or healthy bleeding tissue is reached. A completely healed wound has complete epithelialization (William et al., 2017).
Direct measurement of volume (Depth of wound) | 8 weeks
  Direct measurement of volume using physiological saline:
  The wound will be covered with a sterile polyurethane film and then filled up with physiological saline injected using a needle that pierces the film. The quantity of saline corresponds to the wound volume. Wound volume measurements will be taken at baseline, after 4 weeks (midpoint) and after 8 weeks (HUMBERT et al., 2004).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt